CLINICAL TRIAL: NCT01555827
Title: Retinal Neurodegenerative Signs in Alzheimer's Diseases
Acronym: SIGNAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX2011/19
Record Dates: First submitted 2012-03-14; First posted 2012-03-15 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Alzheimer's Disease
Keywords: Retina; ALzheimer's disease; neurodegenerative signs
MeSH Terms: conditions — Alzheimer Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alzheimer Disease (Experimental)
  Interventions: Other: Ophthalmological examination & Questionnaire
- Control (Active Comparator)
  Interventions: Other: Ophthalmological examination & Questionnaire

INTERVENTIONS:
Other: Ophthalmological examination & Questionnaire — The following examinations will be performed, after pupil dilation:
  * Examination with SD-OCT (macular scans, macular volume, peri-papillary scan, retinal autofluorescence, infer-red and red-free imaging)
  * Colour photographs of the retinal, centered on the macula and on the optic nerve (digital non mydriatic retinal camera)
  * Wide-field colour and autofluorescence imaging (Optomap)
  * Measure of intra-ocular pressure (pneumotonometer)
  The following informations will be collected through a standardized questionnaire, administered face-to-face during the inclusion visit, or at the moment of the verification of eligibility criteria:
  * Age, gender
  * educational level
  * smoking
  * cardiovascular diseases, current medications
  * scores at neuropsychological tests

SUMMARY:
A few studies suggest that patients suffering from neurodegenerative diseases (such a multiple sclerosis or Alzheimer's disease (AD)) show decreased thickness of the retinal nerve fiber layer (RNFL), indicating axonal degeneration. High-definition spectral domain optical coherence tomography (SD-OCT), performed without radiation in a few seconds per eye, offers a precise and standardized estimation of this parameter, which could constitute a biomarker for cerebral axonal degeneration. These RNFL deficits might even be the earliest sign of AD, prior to damage of the hippocampal region that impacts memory.

Besides, some associations of AD with some degenerative diseases of the eye (glaucoma, microvascular abnormalities, age-related macular degeneration (AMD)) have also been reported.

It therefore seems interesting to determine whether RNFL thickness, and other ocular parameters, may give some indications for a better detection of AD and cognitive decline in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for AD cases:
* Diagnosis of probable AD, defined according to the NINCDS-ARDRA criteria51
* Light to moderate severity of the disease, defined by a MMSE score >10 (global evaluation of cognition)
* Patient aged 50 years or more
* Patient benefiting from social insurance

Inclusion criteria for controls:

* Absence of suspicion of dementia, based on normal performance according to age and educational level at neuropsychological testing defined as:
* Free recall ≥17 and total recall ≥40 for the Free and Cued Selective Reminding Test (Grober and Buschke test 52) MMSE ≥ norm for age and educational level (defined by mean - 1 SD)
* Isaac's set test ≥ norm for age and educational level (defined by mean - 1 SD)
* Matched to age and gender of the cases
* Patient benefiting from social insurance

Exclusion Criteria:

Exclusion criteria for all patients :

* History of Parkinson's disease or other neurodegenerative disorder
* History of Horton's disease
* History of inflammatory neuropathies (in particular Devic's disease, multiple sclerosis)
* History of vascular ischemic neuropathies and chronic intracranial hypertension
* History of pituitary tumors
* Presence of diseases (systemic and/or ocular diseases) or behavioural or cognitive symptoms incompatible with eye examination
* Known diabetes
* Person under tutorship or curatorship, person unable to express consent

Additional exclusion criteria for AD cases:

* Dementia of other cause than AD
* Severe AD, defined by MMSE score ≤ 10

Additional exclusion criteria for controls:

* Presence of dementia, of whatever cause

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-03-12 (Actual); Primary Completion 2014-06-07 (Actual); Study Completion 2014-06-07 (Actual)

PRIMARY OUTCOMES:
RNFL thickness measured on a peri-papillary scan of SD-OCT examination. | inclusion visit (day0)

SECONDARY OUTCOMES:
Glaucomatous optic nerve damage observed on colour photographs (cup/disc ratio) | inclusion visit (day0)
Retinal microvascular abnormalities (microaneurysms, micro-hemorrhage, cotton wool spots, arteriovenous nicking), observed on retinal colour photography | inclusion visit (day0)
Macular abnormalities observed on retinal colour photographs (drusen, pigmentary abnormalities, neovascular AMD, atrophic AMD, other retinal diseases) | inclusion visit (day0)
Macular abnormalities observed on macular scans in SD-OCT (drusen, pigmentary abnormalities, neovascular AMD, atrophic AMD, epiretinal membranes, other retinal diseases). | inclusion visit (day0)
Macular abnormalities observed in autofluorescence imaging (increased autofluorescence, decreased autofluorescence, reticular drusen, atrophic AMD, other abnormalities) | inclusion visit (day0)
Macular and peripheral abnormalities diagnosed in wide-field retinal imaging | inclusion visit (day0)
Retinal blood flow velocity (RFI) | inclusion visit (day0)
Intraocular pressure | inclusion visit (day0)
axial length | inclusion visit (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François KOROBELNIK, Pr, Principal Investigator — University Hospital, Bordeaux, France; Delcourt Cécile, Dr, Study Chair — ISPED, bordeaux, France
Locations (1):
- CHU Bordeaux - hôpital Pellegrin, Bordeaux, France